CLINICAL TRIAL: NCT02171221
Title: A Phase I Study of Once-Daily Oral DFP-11207 in Patients With Solid Tumors
Brief Title: Phase I Study of Oral DFP-11207 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Delta-Fly Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D13-11038
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Solid Tumors; Cancer
Keywords: Refractory or relapsed tumors; Antimetabolites, Antineoplastic; Fluorouracil
MeSH Terms: conditions — Neoplasms | interventions — DFP-11207

ARMS (1):
- Oral DFP-11207 (Experimental): DFP-11207: daily oral dosing, 28 day treatment cycle
  Interventions: Drug: Oral DFP-11207

INTERVENTIONS:
Drug: Oral DFP-11207

SUMMARY:
This is a first-in-human, open label, single arm, sequential dose escalation and expansion study of oral DFP-11207 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The Phase I dose escalation portion of the study has been completed. The maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) has been determined. The study will now evaluate the effect of food on the pharmacokinetics of DFP-11207.

The food effect study is a two-step, two-way crossover design to evaluate the pharmacokinetics and bioavailability of oral DFP-11207 capsules. During Cycle 1, oral DFP-11207 capsules are to be taken daily (as a single dose or twice-daily [approximately 12 hours apart]) under fed/fasted conditions. After Cycle 1, the food effect study will be completed and patients will continue to take oral DFP-11207 capsules twice-daily (approximately 12 hours apart) for 28 days of a 28-day treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically-confirmed solid tumors, refractory after standard therapy for the disease or for which conventional systemic chemotherapy is not reliably effective or no effective therapy is available.
2. Aged ≥ 18 years.
3. ECOG Performance Status of 0 or 1.
4. Adequate clinical laboratory values defined as:

   * absolute neutrophil count ≥ 1.5 x 10^9/L
   * platelets ≥ 100 x 10^9/L
   * plasma creatinine ≤ 1.5 x upper limit of normal (ULN) for the institution
   * bilirubin ≤ 1.5 x ULN
   * alanine transaminase (ALT) and aspartate transaminase (AST) < 2.5 x ULN (< 5 x ULN if documented hepatic metastases)
5. Absence of uncontrolled intercurrent illnesses, including uncontrolled infections, cardiac conditions, or other organ dysfunctions.
6. Patients may have measurable or non-measurable disease as defined by RECIST 1.1.
7. Signed informed consent prior to the start of any study specific procedures.
8. Women of child-bearing potential must have a negative serum or urine pregnancy test. Male and female patients must agree to use acceptable contraceptive methods for the duration of the study and for at least one month after the last drug administration.

Exclusion Criteria:

1. Known allergy to fluoropyrimidines or known dihydropyrimidine dehydrogenase (DPD) deficiency.
2. Patients will be excluded if they have received previous chemotherapy, immunotherapy, radiotherapy or any other investigational therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or 5 half-lives for non-cytotoxic agents prior to this study entry.
3. Extensive prior radiotherapy, more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation.
4. Any concomitant condition that in the opinion of the Investigator could compromise the objectives of this study and the patient's compliance.
5. Pregnant or lactating individuals.
6. Current malignancies of another type, with the exception of adequately treated in situ cervical cancer, squamous cell and basal cell skin cancer or other malignancies with no evidence of disease for 2 years or more.
7. Known history of HIV, HBV or HCV infection.
8. Documented or known bleeding disorder.
9. Requirement for anticoagulation treatment that increases international normalized ratio (INR) or activated partial thromboplastin time (aPTT) above the normal range (low dose deep vein thrombosis (DVT) or line prophylaxis is allowed).
10. Clinically evident central nervous system metastases or leptomeningeal disease not controlled by prior surgery or radiotherapy; history of seizure disorder not controlled by anti-seizure medication at the time of enrollment.
11. Cardiac dysfunction defined as myocardial infarction within 6 months of study entry, New York Heart Association Class III or IV heart failure, uncontrolled dysrhythmias or poorly controlled angina.
12. History of serious ventricular arrhythmia (VT or VF, ≥ 3 beats in a row), QTc ≥ 450 msec for men and 470 msec for women, or LVEF ≤ 40% by MUGA or ECHO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-06; Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and to evaluate the safety and tolerability of daily oral dosing of DFP-11207 in patients with solid tumors | Continuous starting on day of first dose (Day 1) up to 30 days after last dose
  The MTD and tolerability will be based on the incidence of adverse events and dose-limiting toxicities in patients. CTCAE 4.0 will be used to grade the severity of adverse events.
For food effect study: To assess PK profiles of DFP-11207 under fed and fasted conditions | Cycle 1, Day 1: pre dose, 4, 10, 24, and 48 hrs post-dose; Day 14: 2, 10 and 24 hrs post-dose; Day 16: pre-dose, 4, 10, and 24 hrs post-dose; Day 18: pre-dose; Day 23: 2 hrs post-dose; Day 29: 2 and 24 hrs post-dose. Cycle 2, Day 1: pre-dose
  Plasma concentration and time data of DFP-11207 metabolites for the food effect study will be determined.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): To measure plasma and urine concentrations of DFP-11207 and its metabolites | Cycle 1, Day 1: 1, 2, 4, 8, 12, 24 and 48 hours post-dose; and on Days 15 and 29
  PK parameters to be measured include area under the concentration curve versus time (AUC) and maximum drug concentration (Cmax)
To determine preliminary efficacy (overall response rate) in solid tumor patients receiving oral DFP-11207 | Every 8 weeks (2 months)
  Response to treatment will be assessed per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ajani JA, Javle M, Eng C, Fogelman D, Smith J, Anderson B, Zhang C, Iizuka K. Phase I study of DFP-11207, a novel oral fluoropyrimidine with reasonable AUC and low Cmax and improved tolerability, in patients with solid tumors. Invest New Drugs. 2020 Dec;38(6):1763-1773. doi: 10.1007/s10637-020-00939-w. Epub 2020 May 6. PMID 32377978